CLINICAL TRIAL: NCT01195506
Title: Study the Novel Functions and Molecular Mechanisms of Vascular Endothelial Growth Factor-C (VEGF-C) in Acute Myeloid Leukemia (AML)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ming-Hsien Chien/stem cell research center, Taipei Medical University
Other Study IDs: 99025
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: We Will Collect the Bone Marrow Specimens From AML Patients
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Vascular endothelial growth factor (VEGF)-C is recognized as a tumor lymphangiogenic factor based on the effects of activated VEGFR3 on lymphatic endothelial cells. VEGFR3 has been proposed as a specific marker for lymphatic endothelial cells. Recent studies indicated that VEGFR3 also expressed in a variety of human malignancies, including lung, colon rectal, or head and neck cancer. Moreover, VEGF-C/VEGFR3 axis was demonstrated in regulating angiogenesis, cell invasion, and metastasis in several solid tumors. The promotion of cell mobility in response to VEGF-C was required the involvement of adhesion molecule contactin-1. In addition to solid tumors, it has been reported that the VEGF-C/VEGFR3 axis is activated in subsets of leukemia patients. Until now, it has been demonstrated that higher endogenous VEGFC levels of acute myelogenous leukemia (AML) cells are related to decreased in vitro and in vivo responsiveness to chemotherapy; an effect that may result from inhibition of apoptosis by increasing Bcl-2/Bax ratios by the VEGF-C/VEGFR3 pathway. Thus, a functional VEGF-C/VEGFR3 system may exist in leukemia. However, the detail information concerning the role of VEGF-C/VEGFR3 in non-solid tumors is still lacking. Bone marrow neoangiogenesis plays a crucial pathogenic and possible prognostic role in AML. The VEGF-C/VEGFR3 axis has been proven in the regulation of solid tumors angiogenesis. In the investigators preliminary study, the investigators found VEGF-C may play a critical role in angiogenesis regulation of leukemic cells by upregulating cyclooxygenase-2 (COX-2). Furthermore, the investigators found that the upregulation of COX-2 also correlate with the VEGF-C-induced proliferation in leukemic cells and this phenomenon might further regulate the chemoresistance of VEGF-C. In this study, the investigators will investigate the extent of angiogenesis and chemoresistance induced by VEGF-C in leukemic cells. This study will provide evidences on the subject of the novel role of VEGF-C in leukemia. With progress in molecular biology of VEGF-C, its value as a therapeutic target is highly promising.

ELIGIBILITY:
Inclusion Criteria:

* patients who were diagnosed acute myeloid leukemia

Exclusion Criteria:

* patients who were diagnosed other type leukemia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients who were diagnosed acute myeloid leukemia
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-09

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hsien Chien, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan